CLINICAL TRIAL: NCT05707208
Title: A Randomized, Controlled Phase II Study of Repeat Dose ST-01 (Lidocaine Polymer Solution) vs Lidocaine for Spermatic Cord Block in Men With Chronic Scrotal Content Pain
Brief Title: A Randomized, Controlled Study of Repeat Dose Sustained Release Lidocaine for Treatment of Chronic Scrotal Pain
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sustained Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ST-CP-202
Record Dates: First submitted 2023-01-20; First posted 2023-01-31 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Chronic Pain
Keywords: Chronic Scrotal Content Pain; Chronic testicular pain; Chronic scrotal pain; Orchialgia; spermatic cord
MeSH Terms: conditions — Chronic Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blind. Participant will not know what study arm they have been randomized to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ST-01 70 mg/mL (Experimental)
  Interventions: Drug: ST-01
- ST-01 140 mg/mL (Experimental)
  Interventions: Drug: ST-01
- 1% Lidocaine HCL (Active Comparator)
  Interventions: Drug: 1% Lidocaine HCL

INTERVENTIONS:
Drug: ST-01 — A sustained release lidocaine formulation designed for the treatment of acute and chronic pain.
  Arms: ST-01 140 mg/mL; ST-01 70 mg/mL
Drug: 1% Lidocaine HCL — Currently approved lidocaine
  Arms: 1% Lidocaine HCL

SUMMARY:
This multi-center, phase 2, randomized, single-blind, three-arm, active-controlled study is comparing repeat doses, every 28 days, of standard of care (SOC) plus ST-01 against SOC plus 1% lidocaine HCL in men experiencing chronic scrotal content pain (CSCP). The main purpose of this study is to determine if repeat injections of ST-01 are safe and effective in reducing pain. After completing a screening phase participants will be randomized into one of three groups: 1) ST-01 70 mg/mL arm, 2) ST-01 140 mg/mL arm, 3) 1% Lidocaine HCL arm (Control). Participants may receive up to 4 study treatment injections given at a minimum of 28-day intervals. Participants randomized to the Control arm will be given the opportunity to cross over to an ST-01 treatment arm after 2 study treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥ 19 years) male
2. Unilateral or bilateral scrotal pain lasting > 3 months
3. Have nociceptive scrotal pain
4. Average daily maximum scrotal pain score over 7 days ≥ 4 on the 0-10 NRS (Appendix 2). Participants with bilateral scrotal pain must be able to distinguish one side with pain score ≥ 4 and the opposite side must have a maximum scrotal pain score of ≤ 3.0 at baseline.
5. Positive response to test spermatic cord block with 1% lidocaine (Lidocaine Hydrochloride Injection, USP, 1%, 10 mg/mL), defined as a decrease in pain score of at least 2 within 1 hour of injection
6. Baseline blood levels without clinically significant abnormalities including liver function tests (alanine aminotransferase [ALT], aspartate aminotransferase [AST], gamma-glutamyl transferase [GGT], and alkaline phosphatase [ALP]) no greater than 50% above the upper limit of normal
7. If sexually active, is willing to use adequate birth control methods to prevent pregnancy over the course of the study

Exclusion Criteria:

1. Negative response to test spermatic cord block, defined as absence of a decrease in pain score of at least 2 within an hour of injection
2. Other pain generator site with NRS pain score ≥ 4 that interferes with evaluation of scrotal pain
3. History of allergic reaction to lidocaine or any component of ST-01
4. Any contraindication to local anesthesia with lidocaine (e.g., known hypersensitivity to anesthetics of the amide type; hypokalemia, complete heart block, anticoagulants (aspirin permitted), antiarrhythmic medication.)
5. Active infection involving the urinary tract or scrotum
6. Inability to give consent
7. Inability to follow up according to the protocol
8. Negative response to previous spermatic cord block
9. Any other condition that the investigator believes may interfere with the safety of the participant, study conduct, or interpretation of the data.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2025-12-04 (Estimated); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Pain Scores on the Numerical Rating Scale (NRS) at 56 days. | 28 days after the second injection of ST-01 or 56 days after the first injection if only one study injection is received.
  To evaluate the change of pain score from baseline to day 56 in the active treatment cohorts (after 1 or 2 injections of ST-01) and compare to the standard of care control group. Pain score being used is the participant reported NRS scale (measured from 0-10 where 0 is no pain and 10 is maximum pain.)

CONTACTS AND LOCATIONS:
Overall Officials: Graeme Boniface, PhD., Study Director — Sustained Therapeutics Inc.
Locations (8):
- Canada (8):
  - Prostate Cancer Centre - Rockyview Hospital, Calgary, Alberta
  - Kelowna General Hospital Clinical Research Department, Kelowna, British Columbia
  - Vancouver Prostate Centre, Vancouver, British Columbia
  - Men's Health Clinic Manitoba, Winnipeg, Manitoba
  - Jonathan Giddens Medicine Professional Corporation, Brampton, Ontario
  - The Fe/Male Health Centre, Oakville, Ontario
  - Mount Sinai Hospital - Men's Health Institute, Toronto, Ontario
  - THEO Medical, Montreal, Quebec